CLINICAL TRIAL: NCT01880099
Title: Cholinergic Enhancement as a Treatment for Nicotine Addiction
Brief Title: A Study to Help People Quit Smoking.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1306012154; 1R21DA034815-01A1 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Nicotine Dependence
Keywords: addiction; smoking; tobacco; cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive; Smoking | interventions — Sugars; Galantamine; Cholinesterase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): Placebo (sugar Pill) will be given daily for 7 weeks.
  Interventions: Drug: placebo
- galantamine 8mg (Active Comparator): Galantamine extended release (8mg) will be given daily for 7 weeks.
  Interventions: Drug: Galantamine 8mg
- Galantamine 16mg (Active Comparator): Galantamine extended release (16mg) will be given daily for 5 weeks starting at week 3 after a two week titration with 8mg galantamine.
  Interventions: Drug: Galantamine 16mg

INTERVENTIONS:
Drug: placebo — placebo compared to 8mg of Galantamine
  Other Names: sugar pill
  Arms: placebo
Drug: Galantamine 8mg — 8mg of galantamine compared to placebo
  Other Names: Acetylcholinesterase inhibitors, Galantamine ER,; Razadyne, Razadyne ER, Reminyl
  Arms: galantamine 8mg
Drug: Galantamine 16mg — 16mg of galantamine compared to placebo
  Other Names: Acetylcholinesterase inhibitors, Galantamine ER,; Razadyne, Razadyne ER, Reminyl
  Arms: Galantamine 16mg

SUMMARY:
You are invited to participate in a research study at the VA Connecticut Healthcare System (West Haven campus) that examines whether a medication called galantamine can improve your learning and memory, and also help you to quit smoking. You have been invited to participate because you currently smoke cigarettes, and want to quit smoking. If you are eligible and agree to be in the study, your participation will last for approximately 8 weeks. To determine if galantamine (8 or 16 mg) is superior to placebo a) in reducing smoking self-administration in a human laboratory model and b) improving abstinence rates at the end of 4 weeks of treatment.

DETAILED DESCRIPTION:
We propose a double-blind, placebo-controlled, outpatient study with a between-groups design. Seventy-two male and female smokers will be randomly assigned to one of the 3 treatment conditions: GAL (8 or 16 mg/day) or placebo. The dose of GAL will be gradually increased to the target doses over a 2-week period (Table 2). During Week 3, following overnight abstinence from smoking, participants will present for a laboratory Test Session in which they will have the option of cigarette self-administration. After this Test Session is completed, smokers will be maintained on their randomized medication condition for an additional 4-week period. Smokers will establish a quit date at the beginning of this Treatment Phase, and will receive brief weekly behavioral treatment for the 4 weeks of this phase. Additionally, at the beginning of Week 3, participants will be given a PDA that will administer EMA assessments. The study medication will be tapered after the end of Week 4 of the Treatment Phase. Participants will be contacted by phone at one week, and one month, after treatment termination to inquire about any adverse events and about their recent smoking status.

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 55 years;
* history of smoking daily for the past 12 months, at least 10 cigarettes daily;
* in good health as verified by medical history, screening examination, and screening laboratory tests;
* for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* History of GAL allergy;
* requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history (in the past 6 months);
* serious medical illness including asthma, diabetes, bradycardia, or other arrhythmias and major cardiovascular, renal, endocrine, or hepatic disorders;
* abuse of alcohol or any other illicit or prescription drugs;
* use of any other tobacco products, including smokeless tobacco and nicotine products; and
* inability to fulfill all scheduled visits and examination procedures throughout the study period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Veteran Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (sugar Pill) will be given daily for 7 weeks.
  placebo: placebo compared to 8mg of galatamine
- Galantamine 8mg: Galantamine extended release (8mg) will be given daily for 7 weeks.
  Galantamine 8mg: 8mg of galatamine compared to placebo
- Galantamine 16mg: Galantamine extended release (16mg) will be given daily for 5 weeks starting at week 3 after a two week titration with 8mg galantamine.
  Galantamine 16mg: 16mg of galatamine compared to placebo
Period: Overall Study
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
Started | 17 | 21 | 22
Completed | 9 | 11 | 15
Not Completed | 8 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg | Total
Number analyzed (Participants) | 17 | 21 | 22 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 22 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 10 | 24
  Male | 11 | 13 | 12 | 36
Region of Enrollment [Number; unit: participants]
  United States | 17 | 21 | 22 | 60

OUTCOME MEASURES:

1. Primary Outcome: Smoking Choice Procedure
Description: After overnight abstinence, participants will receive 10 tokens at the beginning of the smoking choice session. These tokens can be exchanged for money (0.75$ / token) or 2 cigarette puffs. The session starts with sample smoking of 2 puffs that allows subjective responses to me measured after abstinence. 15 min later, participants make their first choice, followed by 9 additional choices, every 15 minutes.
Time Frame: Data was acquired during a single test session during week 3 of drug intervention.
Population: The number of participants analyzed per arm for this outcome is different than participant flow data because not every participant completed the smoking choice session.
Measure: Mean (Standard Deviation); unit: # of choices to smoke (out of 10)
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
Number analyzed (Participants) | 13 | 15 | 20
# of choices to smoke (out of 10) | 3.00 (3.08) | 1.00 (1.00) | 0.85 (1.35)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 8/17 | 13/21 | 11/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Galantamine 8mg (N=21) | Galantamine 16mg (N=22)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (5)
Vomitting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Constipation (General disorders) | 2 (2) | 2 (2) | 3 (3)
Loss of Appetite (General disorders) | 4 (4) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2)
Nervousness (Psychiatric disorders) | 4 (4) | 4 (4) | 5 (5)
Restlessness (Psychiatric disorders) | 3 (3) | 6 (6) | 5 (5)
Difficulty sleeping (General disorders) | 2 (2) | 5 (5) | 8 (8)
Drowsy (General disorders) | 1 (1) | 6 (6) | 4 (4)
Fatigue (General disorders) | 2 (2) | 5 (5) | 3 (3)
Anger (General disorders) | 2 (2) | 4 (4) | 5 (5)
Depressed mood (Psychiatric disorders) | 2 (2) | 5 (5) | 4 (4)
Confusion (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2)
Teary/dry eyes (General disorders) | 2 (2) | 3 (3) | 5 (5)
Runny nose (General disorders) | 4 (4) | 4 (4) | 3 (3)
Back/ muscle pain (General disorders) | 4 (4) | 4 (4) | 5 (5)
Sweating (General disorders) | 3 (3) | 4 (4) | 2 (2)
Excessive hunger (General disorders) | 2 (2) | 5 (5) | 6 (6)
dry mouth (General disorders) | 1 (1) | 4 (4) | 6 (6)
change in the ability to taste food (General disorders) | 0 (0) | 4 (4) | 3 (3)
heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5)
blurred vision (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
Gas (Gastrointestinal disorders) | 3 (3) | 5 (5) | 3 (3)
lighted headed (General disorders) | 0 (0) | 2 (2) | 2 (2)
weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Sudden hunger (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (5)
concentration (General disorders) | 2 (2) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Aggresive behavior (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
mood swings (General disorders) | 2 (2) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No